CLINICAL TRIAL: NCT05852613
Title: Effect of High Power Laser Therapy on Pain and Electrophysiological Study in Cervical Radiculopathy Patients: Randomized Controlled Trial
Brief Title: Effect of HPLT on Pain and Electrophysiological Study in Cervical Radiculopathy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Ahmed Sherif Sherif, Physiotherapist at Al-Minshawy General Hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dina Ahmed Sherif Sherif
Record Dates: First submitted 2023-04-27; First posted 2023-05-10 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cervical Radiculopathy
Keywords: High power laser therapy; Cervical radiculopathy; Electrophysiological study; nerve conduction study; electromyography
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: The current study will include twenty patients with unilateral cervical radiculopathy caused by disc prolapse at the level of C5 - C6 or C6 - C7. Patients will be diagnosed on the basis of clinical (history and physical examination) and radiological examination (MRI). All subjects will be evaluated using the same procedures.
  - Patients will be randomly assigned into two equal matched groups
  Group (A) study group: (N=10) this group will receive high power laser therapy (HPLT) for 15 minutes in addition to selected physical therapy program (hot pack, US for 5 min, exercise for 20min) for 8 session two times weekly for 4 weeks.
  Group (B) control group: (N=10) this group will receive the same selected physical therapy program only (hot pack,US for 5 min, exercise for 20 min) for 8 session.
  All patients will attended the physical therapy clinic two times weekly for 4 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) (Experimental): this group will receive high power laser therapy (HPLT) for 15 minutes in addition to selected physical therapy program for 8 session two times weekly for 4 weeks.
  Interventions: Device: high power laser therapy (HPLT); Combination Product: selected physical therapy program
- Group (B) (Active Comparator): this group will receive the same selected physical therapy program only for 8 session.
  All patients will attended the physical therapy clinic two times weekly for 4 weeks .
  Interventions: Combination Product: selected physical therapy program

INTERVENTIONS:
Device: high power laser therapy (HPLT) — high power laser therapy (HPLT) will be produced by A LEVELASER EZ1 EASYONE device which produces a Ga Al As CW diode laser with pulsed emission 980 nm and maximum average power 5 W with a high level of energy penetration. While the patient is in a prone position and the head slightly bends to the front, The treatment will be performed at a distance of 60-70 cm, perpendicular to the cervical region, in a pulsed mode of 4 Hz, wavelength = 980 nm, radiation power density P = 4 W in the scan phase and 2 W in the acupuncture phase and energy 840 J. Patients will receive pulsed HPLT laser treatment for 8 minutes. Scanning will be performed transversely and longitudinally to the bilateral paraspinal muscles, inter-scapular area, upper trapezius and the neck region for 6 minutes followed by 2 minutes acupuncture. Protective goggles will be used to prevent direct eye contact of the laser beam.
  Other Names: LEVELASER EZ1 EASYONE device
  Arms: Group (A)
Combination Product: selected physical therapy program — hot pack, US for 5 min, exercise for 20 min.

SUMMARY:
The goal of this clinical trial is :

To determine the effect of high power laser therapy on pain and electrophysiological study in patients with cervical radiculopathy.

The main question it aims to answer :

Is there a significant effect of high power laser therapy (HPLT) on pain and electrophysiological study in patients with cervical radiculopathy?

Twenty patients with cervical radiculopathy caused by disc prolapse at the level of C5 - C6 or C6 - C7 will randomly assigned into two equal matched groups;

* group A (study group) N=10: this group will receive high power laser therapy (HPLT) for 8 minutes in addition to selected physical therapy program
* group B (control group) N=10: this group will receive the same selected physical therapy program only (hot pack, US for 5 min, exercise for 20 min) for 8 session.

All patients will attend the physical therapy clinic two times weekly for 4 weeks.

The evaluation was done by nerve conduction study (NCS) and needle electromyography (EMG) before and after the treatment in addition to visual analogue scale (VAS).

HYPOTHESES:

Null hypothesis: There is no significant effect of high power laser therapy on pain and electrophysiological study in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
This current study will be designed to determine the effect of high power laser therapy on pain and electrophysiological study in patients with cervical radiculopathy. This study will be carried out at outpatient clinic of Faculty of Physical Therapy, Cairo University.

Twenty patients with cervical radiculopathy caused by disc prolapse at the level of C5 - C6 or C6 - C7 cervical radiculopathy will be selected from outpatient clinic of Faculty of Physical Therapy, Cairo University and outpatient clinic of Qasr El- Aini Hospitals.

On approval to participate in the study, all subjects will sign an informed consent form after receiving full information on the purpose of study, procedure, possible benefits, privacy and use of data, and their rights to withdraw from the study whenever they want.

Sample size:

Sample size calculation is performed using G*POWER statistical software (version 3.1.9.2; Franz Faul, Universitat Kiel, Germany) and revealed that the required sample size for this study is N=20.

Statistical analysis

* Descriptive statistics in form of mean, standard deviation and frequency will be conducted for the subject's demographics and collected data.
* Paired samples T Test procedure will be used to compare the means of two variables for a single group.
* Independent sample T Test Procedure will be used to compares means for two groups.
* Pearson Correlation Coefficient will be conducted to determine the correlation between electrophysiological study and pain intensity.
* The level of significance for all statistical tests will be set at p < 0.05.
* All statistical tests will be performed through the statistical package for social studies (SPSS) version 25 for windows. (IBM SPSS, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Twenty patients with unilateral cervical radiculopathy due to disc prolapse at the level of C5 - C6 or C6 - C7.
* Age ranges from 30 to 50 years.
* Patients will be both sexes.
* Patients will be diagnosed by clinical and radiological examination.
* Presence of sensory changes as pain and paresthesia (numbness, tingling, burning) in the upper extremity.
* Pain severity should be moderate or severe.
* Reporting a minimum pain score of 4 on a 10-point Visual Analogue Scale (VAS).
* Duration of pain ranges from (3-12) months.

Exclusion Criteria:

* Diabetic patient.
* Patients with peripheral neuropathy or entrapment syndrome.
* Previous cervical or shoulder surgery.
* Fracture of the bones of upper extremity.
* Major neurological condition (e.g., stroke, multiple sclerosis, Epilepsy, Meningitis, and Brain tumor).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
pain severity | before and after one month of treatment
  using a 0-10 cm visual analog scale (VAS). Patients were asked to make a handwritten mark on a 100 mm line (10cm). This line represents a continuum between no pain or discomfort (zero), to the worst pain (10) that the patient could feel. The measure was taken by a ruler from the starting point of the scale to the mark the patient scored in millimeters.
  The results were interpreted as: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm), (Jensen 2003). Patients should have moderate to severe neck pain to be included in the study. The pain intensity was recorded before and after the study.
F wave | before and after one month of treatment
  for both median and ulnar nerves of both upper extremities

SECONDARY OUTCOMES:
nerve conduction studies (NCS) | before and after one month of treatment
  for both median and ulnar nerves of both upper extremities
electromyography (EMG) | before and after one month of treatment
  using a bipolar needle electrode to biceps brachii, triceps and first dorsal interosseus muscles of both upper extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf A Darwish, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, El Behoth, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barassi G, Supplizi M, Prosperi L, Irace G, Younes A, Della Rovere M, Rabini A, Colombo A, Di Iorio A. Dual-wavelength high-power laser therapy and neuromuscular manual therapy in chronic neck pain: a randomized clinical trial. J Biol Regul Homeost Agents. 2021 Mar-Apr;35(2):767-773. doi: 10.23812/21-37-L. No abstract available. PMID 33902272
- [Background] Alayat MS, Mohamed AA, Helal OF, Khaled OA. Efficacy of high-intensity laser therapy in the treatment of chronic neck pain: a randomized double-blind placebo-control trial. Lasers Med Sci. 2016 May;31(4):687-94. doi: 10.1007/s10103-016-1910-2. Epub 2016 Feb 25. PMID 26914684
- [Background] Venosa M, Romanini E, Padua R, Cerciello S. Comparison of high-intensity laser therapy and combination of ultrasound treatment and transcutaneous nerve stimulation in patients with cervical spondylosis: a randomized controlled trial. Lasers Med Sci. 2019 Jul;34(5):947-953. doi: 10.1007/s10103-018-2682-7. Epub 2018 Nov 15. PMID 30443883
- [Background] Conforti M, Fachinetti GP. High power laser therapy treatment compared to simple segmental physical rehabilitation in whiplash injuries (1 degrees and 2 degrees grade of the Quebec Task Force classification) involving muscles and ligaments. Muscles Ligaments Tendons J. 2013 Jul 9;3(2):106-11. doi: 10.11138/mltj/2013.3.2.106. Print 2013 Apr. PMID 23888293
- [Background] Kenareh R, Mirmohammadi SJ, Khatibi A, Shamsi F, Mehrparvar AH. The Comparison of The Efficacy of Photobiomodulation and Ultrasound in the Treatment of Chronic Non-specific Neck Pain: A Randomized Single-Blind Controlled Trial. J Lasers Med Sci. 2021 May 17;12:e20. doi: 10.34172/jlms.2021.20. eCollection 2021. PMID 34733743